CLINICAL TRIAL: NCT01985009
Title: Evaluating the Diagnosis Accuracy of the Controlled Attenuation Parameter(CAP) Measured by FibroScan® (Either With M+ or XL+ Probe) in Patient With Non-Alcoholic Fatty Liver Disease (NAFLD)Using Liver Biopsy as Reference.
Brief Title: Prospective, Cross-sectional and Multicenter Study, Evaluating the Diagnosis Accuracy of the Controlled Attenuation Parameter(CAP) Measured by FibroScan® (Either With M+ or XL+ Probe) in Patient With Non-Alcoholic Fatty Liver Disease Using Liver Biopsy as Reference.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M118
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2016-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibroscan® (Other): Single arm study. See intervention item for détails..
  Interventions: Device: FibroScan® examination.

INTERVENTIONS:
Device: FibroScan® examination. — The study involves adults' patients with suspected Non-Alcoholic Fatty Liver Disease(NAFLD). The FibroScan® is a device equipped with probes (M+ or XL+), each of which consists of an ultrasonic transducer mounted on the axis of a mechanical vibrator. Liver stiffness and CAP measurements are performed on the right lobe of the liver with the patient in a dorsal decubitus and maximal abduction position. The procedure is non-invasive and painless.

SUMMARY:
The non-alcoholic fatty liver disease (NAFLD) represents the most common cause of liver disease in the western world. It can progress from steatosis to non-alcoholic steatohepatitis (NASH), and then onto cirrhosis where there is a concomitant risk of developing hepatocellular carcinoma (HCC). The prevalence of hepatic steatosis is high, ranging from 16 to 31% in the general population, up to 80% in the obese populationand up to 96% in severely obese patients.

Liver biopsy (LB) has traditionally been regarded as the gold standard for the assessment of patients with NAFLD, although it has several limitations. LB has a potential sampling error, is an invasive and often painful procedure.

The natural history of patients with NAFLD is generally determined by the extent of liver fibrosis, hence non-invasive assessment of fibrosis with FibroScan® is often sufficient. For patients with proven NASH, changes in hepatic steatosis and serum ALT levels may provide information on the patient's course and/or response to treatment.

Several clinical studies have shown the benefit of measuring hepatic stiffness with the FibroScan® machine using the M+ probe. The ability to identify significant fibrosis and cirrhosis has been demonstrated in normal and overweight patients affected with chronic hepatitis B and C, biliary diseases, alcohol related liver disease (ALD) and NAFLD.

Recently, Echosens has also developed a novel ultrasonic controlled attenuation parameter (CAP) designed to quantify hepatic steatosis using a process based on vibration controlled transient elastography (VCTE™). Studies comparing CAP with liver biopsies in multi-aetiology cases and patients with Hepatitis C Virus (HCV) have shown that there is a good correlation between steatosis assessed histologically and using CAP.

The main objective of this prospective study is to evaluate the diagnosis accuracy of the Controlled attenuation Parameter (CAP) measured by FibroScan® (either with M+ or XL+)in patients with NAFLD to assess liver steatosis using biopsy as a reference.

The study involves adults' patients with suspected NAFLD scheduled to have a liver biopsy within 2 weeks of fibroscan examination and followed by the Hepatology service of four centers in United Kingdom.

Approximately 450 patients (of which 350 will be evaluable) will be enrolled in this study: Around 100 patients will be measured with the M+ probe and around 250 with the XL+ probe.

The inclusion period is from 18 to 24 months. Starting date: January 2014. End of recruitment: June 2017. The duration of the study for a patient is from 1 to 7 days, depending to the exams calendar.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Patients must be able to give written informed consent
* Patients with suspected NAFLD
* Patients scheduled to have a liver biopsy within 2 weeks of Fibroscan examination
* HBsAg negative, Anti-HCV negative, HCV-RNA negative, HBV-DNA negative

Exclusion Criteria:

* Unable or unwilling to provide written informed consent
* Patients with ascites
* Pregnant women
* Patients with any active implantable medical device (such as pacemaker or defibrillator)
* Patients who have had a liver transplant
* Patients with cardiac failure and/or significant valvular disease
* Patients with hematochromatosis
* Refusal to undergo a liver biopsy and/or blood test
* Alcohol consumption above recommended limits (>14 units/week for women and >21 units/week for men)
* Confirmed diagnosis of active malignancy, or other terminal disease
* Patient participation in another clinical trial within the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Performance of CAP will be assessed using ROC analysis for the detection of steatosis above 5% - 10% - 30% and 60% using liver biopsy as the reference. | Up to 24 month

SECONDARY OUTCOMES:
Clinical, histological and biological factors associated CAP will be assessed using multivariate correlation. | Up to 24 month

OTHER OUTCOMES:
Performances of stiffness will be assessed by ROC analysis for the diagnosing above or equal to F2 fibrosis and cirrhosis (F4)using liver biopsy as the reference. | Up to 24 month

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Royal Free Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Queen's Medical Centre Nottingham, Nottingham
  - John Radcliffe Hopsital, Oxford
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Newsome PN, Sasso M, Deeks JJ, Paredes A, Boursier J, Chan WK, Yilmaz Y, Czernichow S, Zheng MH, Wong VW, Allison M, Tsochatzis E, Anstee QM, Sheridan DA, Eddowes PJ, Guha IN, Cobbold JF, Paradis V, Bedossa P, Miette V, Fournier-Poizat C, Sandrin L, Harrison SA. FibroScan-AST (FAST) score for the non-invasive identification of patients with non-alcoholic steatohepatitis with significant activity and fibrosis: a prospective derivation and global validation study. Lancet Gastroenterol Hepatol. 2020 Apr;5(4):362-373. doi: 10.1016/S2468-1253(19)30383-8. Epub 2020 Feb 3. PMID 32027858
- [Derived] Eddowes PJ, Sasso M, Allison M, Tsochatzis E, Anstee QM, Sheridan D, Guha IN, Cobbold JF, Deeks JJ, Paradis V, Bedossa P, Newsome PN. Accuracy of FibroScan Controlled Attenuation Parameter and Liver Stiffness Measurement in Assessing Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 May;156(6):1717-1730. doi: 10.1053/j.gastro.2019.01.042. Epub 2019 Jan 25. PMID 30689971